CLINICAL TRIAL: NCT03311594
Title: The Alcohol-Pain Connection: Mechanisms and Genetic/Psychological Correlates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Joseph W. Ditre, Professor, Syracuse University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 5R01AA024844-02 (NIH); 5R01AA024844 (NIH)
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Pain; Alcohol Drinking; Acute Pain; Drinking Behavior
Keywords: Alcohol; Pain
MeSH Terms: conditions — Pain; Alcohol Drinking; Acute Pain; Drinking Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Low Alcohol Consumption and No Pain Induction (Experimental): Condition 1: Low alcohol consumption Condition 2: No pain group
  Interventions: Drug: Low Alcohol; Other: No Pain Induction
- Low Alcohol Consumption and Pain Induction (Experimental): Condition 1: Low alcohol consumption Condition 2: Pain group
  Interventions: Drug: Low Alcohol; Other: Pain Induction
- Moderate Alcohol Consumption and No Pain Induction (Experimental): Condition 1: Moderate alcohol consumption Condition 2: No pain group
  Interventions: Drug: Moderate Alcohol; Other: No Pain Induction
- Moderate Alcohol Consumption and Pain Induction (Experimental): Condition 1: Moderate alcohol consumption Condition 2: Pain group
  Interventions: Drug: Moderate Alcohol; Other: Pain Induction
- Placebo Alcohol Consumption and No Pain Induction (Placebo Comparator): Condition 1: Placebo alcohol consumption Condition 2: No pain group
  Interventions: Drug: Placebo Alcohol; Other: No Pain Induction
- Placebo Alcohol Consumption and Pain Induction (Experimental): Condition 1: Placebo alcohol consumption Condition 2: Pain group
  Interventions: Drug: Placebo Alcohol; Other: Pain Induction
- Control and No Pain Induction (Placebo Comparator): Condition 1: No alcohol consumption Condition 2: No pain group
  Interventions: Other: No Pain Induction
- Control and Pain Induction (Experimental): Condition 1: No alcohol consumption Condition 2: Pain group
  Interventions: Other: Pain Induction

INTERVENTIONS:
Drug: Low Alcohol — Low Alcohol Consumption
  Arms: Low Alcohol Consumption and No Pain Induction; Low Alcohol Consumption and Pain Induction
Drug: Moderate Alcohol — Moderate Alcohol Consumption
  Arms: Moderate Alcohol Consumption and No Pain Induction; Moderate Alcohol Consumption and Pain Induction
Drug: Placebo Alcohol — Placebo Alcohol Consumption
  Arms: Placebo Alcohol Consumption and No Pain Induction; Placebo Alcohol Consumption and Pain Induction
Other: Pain Induction — 10% capsaicin solution placed on forearm and heat induction
  Arms: Control and Pain Induction; Low Alcohol Consumption and Pain Induction; Moderate Alcohol Consumption and Pain Induction; Placebo Alcohol Consumption and Pain Induction
Other: No Pain Induction — Water placed on forearm
  Arms: Control and No Pain Induction; Low Alcohol Consumption and No Pain Induction; Moderate Alcohol Consumption and No Pain Induction; Placebo Alcohol Consumption and No Pain Induction

SUMMARY:
The societal impact of heavy alcohol consumption and chronic pain is substantial and warrants the existing research investment into their etiology and treatment. Moreover, evidence of significant co-occurrence between these conditions offers an opportunity to examine mechanisms in the alcohol-pain connection that may inform the development of novel treatments. Consistent with NIH PA-15-026 (Mechanistic Studies of Pain and Alcohol Dependence), the goal of the proposed study is to examine several complex and potentially bidirectional relations between pain and alcohol in one overarching model, which has never been attempted in a human experimental paradigm. The primary study aims are as follows: (1) to conduct the first test of both pharmacological and expectancy effects in acute alcohol analgesia among humans; (2) to conduct the first test of pain as a proximal antecedent of urge to drink and ad lib alcohol consumption, and to test whether acute analgesic effects predict pain-induced alcohol urge/consumption; (3) to test associations between study outcomes and candidate genetic polymorphisms that have been implicated in pain-alcohol processes; and (4) to conduct exploratory analyses of gender and pain relevant cognitive-affective factors as moderators of these outcomes. Participants will include 280 moderate-to-heavy drinkers recruited from the local community. Experimental methods will include alcohol administration (moderate dose vs. low dose vs. placebo vs. control) and pre/post assessment of static/dynamic pain responses, and capsaicin/heat pain induction (vs. no pain induction) followed by assessment of urge to drink and ad lib alcohol consumption. By employing a novel experimental paradigm, the study results will provide internally valid data with clear and direct implications for translating these findings to clinical applications. It is our expectation that this work will catalyze future research and inform clinical practice by establishing an experimental platform that allows for the demonstration of causal effects, the evaluation of treatment components prior to conducting costly clinical trials, and the identification of important theory-based biopsychosocial mechanisms that can inform the development of novel integrated treatments for individuals with co-occurring pain and alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

1. be 21-64 years of age
2. be classified as a moderate or heavy drinker based on the Quantity-Frequency-Variability Questionnaire, which will assure that participants currently (last 3 months) consume alcohol in amounts similar to what will be administered or available in the proposed experiments

Exclusion Criteria:

1. current acute or chronic pain
2. chili pepper allergies (contraindicated for capsaicin)
3. current use of prescription pain medications
4. any possibility of being pregnant (verified at session via a pregnancy test)
5. self-reported history of or treatment for psychiatric or alcohol/other drug problems
6. participants who are under the age of 21 or who do not have a government issued ID; and
7. medical conditions that contraindicate the use of alcohol (e.g., diabetes, liver disease).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 379 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Alcohol Urge/Consumption | 15 minutes
  Amount of alcohol consumed and self-reported urge to drink
Pain Response | 40 minutes
  Pain Quantitative Sensory Testing before and after beverage consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ditre JW, LaRowe LR, Powers JM, White KM, Paladino MB, Zvolensky MJ, Glatt S, Maisto SA. Pain as a causal motivator of alcohol consumption: Associations with gender and race. J Psychopathol Clin Sci. 2023 Jan;132(1):101-109. doi: 10.1037/abn0000792. Epub 2022 Dec 8. PMID 36480413